CLINICAL TRIAL: NCT04340089
Title: The Effect of Squatting on the Toilet on Gastric Transit Time and Complete Examination Rate of Capsule Endoscopy
Brief Title: Squatting on the Toilet and Capsule Endoscopy
Acronym: SC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: wuzhixuan2003
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Intestinal Diseases
Keywords: squatting on the toilet; capsule endoscopy
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observation group: the patients can go to squatting on the toilet at any time as they want to after taking the capsule
  Interventions: Behavioral: squatting on the toilet
- control group: The patients can move freely

INTERVENTIONS:
Behavioral: squatting on the toilet — the patients could go to squatting on the toilet at any time as they want to after taking the capsule
  Groups: observation group

SUMMARY:
This study evaluates the effect of squatting on the toilet on gastric transit time and complete examination rate of capsule endoscopy.In the observation group, the patients could go to squatting on the toilet at any time as they want to after taking the capsule.

DETAILED DESCRIPTION:
The subjects were divided into a control group and an observation group according to whether the patient squatted in the toilet, In the control group, the patients took discontinuous right lateral position, walked on a flat road and climbed the stairs alternately. In the observation group, in addition to the above ways, the patients could go to squatting on the toilet at any time in the first hour after taking the capsule. The operator observed the position of capsule every one hour. The examination was over when capsule endoscopy entered the colon. If the capsule remained in the small intestine, the examination continued until the capsule ran out of power.

ELIGIBILITY:
Inclusion Criteria:

* unexplained gastrointestinal bleeding, unexplained chronic abdominal pain and diarrhea, suspected Crohn's disease, suspected small intestinal tumor, and patients needing to exclude small intestinal diseases.

Exclusion Criteria:

* suspected intestinal obstruction and intestinal stenosis, esophageal stenosis or dysphagia, history of abdominal operation, or diabetes mellitus.

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: the patients needed to the examination of capsule endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
CER | 72 hours
  complete examination rate

SECONDARY OUTCOMES:
GTT | 72 hours
  gastric transit time

CONTACTS AND LOCATIONS:
Overall Officials: Song He, Dr., Principal Investigator — Director of department
Locations (1):
- The second affiliated hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided